CLINICAL TRIAL: NCT05695794
Title: Evaluation of the Effect of Different Bed Head Heights After Rhinoplasty on Edema, Ecchymosis, Respiratory Function and Sleep Quality
Brief Title: The Effect of Different Bed Head Heights on Patients After Rhinoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Şevval Polat, Principal Investigator, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BartınU-SBF-SP-01
Record Dates: First submitted 2022-11-22; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Rhinoplasty
Keywords: Rhinoplasty; Edema; Ecchymosis; Respiratory Function Tests; Sleep Quality
MeSH Terms: conditions — Edema; Ecchymosis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: experimental group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group with a bed head height of 45 degrees (Other): The bed head height of the patients in this group will be adjusted to 45 degrees. This group was determined as the control group since the patients were given a 45-degree head height as a standard in the hospital where the study would be conducted.
  Interventions: Other: the group with a bed head height of 45 degrees
- the group with a bed head height of 30 degrees (Experimental): The bed head height of the patients in this group will be adjusted to 30 degrees. This group was determined as the experimental group since the patients were given a 45-degree head height as a standard in the hospital where the study would be conducted.
  Interventions: Other: the group with a bed head height of 30 degrees

INTERVENTIONS:
Other: the group with a bed head height of 45 degrees — Edema, ecchymosis, respiratory function and sleep quality will be evaluated by giving a 45 degree head height to 30 patients determined by Randomizer.org.
  Other Names: Nursing care intervention for positioning appropriately after surgery
  Arms: the group with a bed head height of 45 degrees
Other: the group with a bed head height of 30 degrees — Edema, ecchymosis, respiratory function and sleep quality will be evaluated by giving 30 degrees of bed head height to 30 patients determined by Randomizer.org.
  Other Names: Nursing care intervention for positioning appropriately after surgery
  Arms: the group with a bed head height of 30 degrees

SUMMARY:
This study will be conducted to evaluate the effect of different bed head heights (thirty degrees and forty-five degrees) given to patients after rhinoplasty surgery on periorbital edema, periorbital ecchymosis, respiratory function and sleep quality.

DETAILED DESCRIPTION:
The nose is morphologically a functional and aesthetic organ. These two concepts are inseparable and interact with each other. The nose is one of the structures most exposed to trauma, especially on the face. Rhinoplasty is one of the most common operations performed by plastic surgeons for functional correction or cosmetic purposes. When we examine the history of nose surgeries, we see that nose surgeries begin with reconstruction. Reduction rhinoplasty emerged later and forms the basis of today's rhinoplasty. The treatment of nasal trauma was first mentioned in the Edwin Smith Surgical Papyrus in 3000 BC (BC). In these papyri, 48 patients were reported to have been treated surgically. In the 5th century BC, Hippocrates made detailed patient analysis in his work named "Mochlicon" and classified nasal injuries from simple fracture to complicated. He discussed the reduction of nasal bones and their treatment with poultice. Most historians reported that nasal reconstruction was first mentioned in Sanskrit writings in Ancient India. In these writings, it was reported that the noses of Hindu women were cut as punishment. B.C. In the 6th century; Sushruta performed the reconstruction of the nose using his own instruments. He performed tissue transfer from forehead and cheek to nose. He called it the Indian Method. Sushruta mentioned the nasal reconstruction methods he developed in his book Samhita. 1st century There are articles describing the nose reconstruction in the book called De Medicina, which was written in Rome. VII. In the sculpture of the Byzantine Emperor in the 16th century, it is depicted that there is a scar on his forehead. It was accepted that this was a sign of nasal reconstruction. With the Muslim conquest of India, the nose reconstruction techniques applied in India started to be used in Muslim countries as well. XIV. Since the 19th century, the development of nose surgery has accelerated in Europe. XIV. Since the 19th century, the development of nose surgery has accelerated in Europe. XV. In the 19th century, the Italian surgeon Branca introduced the Indian Method in nose surgery to Europe. Branca's son Antonio, on the other hand, developed a new method in nose surgery and named it the "Italian Method". Nose surgeries have been performed with open technique for centuries. It was Jacques Joseph who coined the term "open rhinoplasty" for the first time, which he would later adopt in Millard and Gillies. Joseph is the scientist who introduced techniques such as nasal dorsum reconstruction with bone grafting and cartilage suturing to rhinoplasty. The first to describe the closed approach in rhinoplasty was John O Roe (1887), an American surgeon. Later, Weir presented the closed technique in 1892 and the German J. Joseph in 1898. In the closed technique, incisions are made through the nose, and in the open technique, a very small incision of approximately 2 millimeters in length is made in the columella of the nose (the part visible from the outside of the middle support) in addition to the incisions made through the nose. If the nose wings need to be narrowed; Additional incisions of approximately 5-6 millimeters can also be made so that they remain in the fold at the base of the nose wings. As with all surgical interventions, the comfort of the patient is important after rhinoplasty. Factors affecting the comfort of the patient in the early period after rhinoplasty; nausea, vomiting, bleeding, periorbital edema, periorbital ecchymosis, nasal airway obstruction and pain. Among these, the factors that most affect the comfort of the patient are; pain, periorbital edema and periorbital ecchymosis. Occurrence of periorbital edema and periorbital ecchymosis; Even if it is a natural result of the procedure, it is an undesirable result for patients who undergo this procedure with aesthetic demands. Postoperative periorbital edema and periorbital ecchymosis cause a delay in patients' return to daily life and adversely affect their social lives. Depending on the degree of periorbital edema, visual difficulties may also be experienced in the early postoperative period. Periorbital ecchymosis occurs by extravasation from damaged vessels and can be positioned by the effect of gravity. This may cause color change in the operation area and delays in returning to the patient's normal social life. Various agents such as corticosteroids, arnica, lidocaine, adrenaline combination and Melilotus extract and cold application methods for different durations have been used to reduce periorbital edema and periorbital ecchymosis after rhinoplasty. In line with these scanned literatures, it was observed that studies on bed head height after rhinoplasty were limited, and it was observed that there was no common decision on bed head heights given to patients in practice.For these reasons, it was decided to examine the effect of different bed head heights (thirty degrees and forty-five degrees) given to patients on periorbital edema, periorbital ecchymosis and respiratory functions.

ELIGIBILITY:
Inclusion Criteria:

* Participating in the research voluntarily
* Patients over the age of 18
* Patients who have undergone rhinoplasty for aesthetic purposes
* Can speak Turkish
* Patients who do not have a mental disability that may interfere with communication
* Patients who had rhinoplasty with open technique
* Patients without diagnosed respiratory and sleep disorders

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients under the age of 18
* Patients who underwent rhinoplasty surgery due to trauma
* Patients with mental disabilities who interfere with communication
* Patients who cannot adapt to bed height
* Patients who had rhinoplasty surgery with the closed technique
* Patients with diagnosed respiratory and sleep disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-03-21 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Periorbital edema score | 1 hour after surgery
  This measurement tool has a single question and has options that score between 0-4:
  0 points: No periorbital edema
  1. point: Mild periorbital edema
  2. points: Periorbital edema enlarged towards the iris layer of the eye
  3. points: Periorbital edema covering the iris
  4. points: Severe periorbital edema covering the eyelid completely With this measurement tool, the periorbital edema status of all patients will be evaluated in terms of periorbital edema as stated above, and a score will be given by the researcher immediately after the patients come to the service from the operating room, at the 1st hour, 4th hour and 24th hour.
Periorbital edema score | 4 hours after surgery
  This measurement tool has a single question and has options that score between 0-4:
  0 points: No periorbital edema
  1. point: Mild periorbital edema
  2. points: Periorbital edema enlarged towards the iris layer of the eye
  3. points: Periorbital edema covering the iris
  4. points: Severe periorbital edema covering the eyelid completely With this measurement tool, the periorbital edema status of all patients will be evaluated in terms of periorbital edema as stated above, and a score will be given by the researcher immediately after the patients come to the service from the operating room, at the 1st hour, 4th hour and 24th hour.
Periorbital edema score | 24th hour after surgery
  This measurement tool has a single question and has options that score between 0-4:
  0 points: No periorbital edema
  1. point: Mild periorbital edema
  2. points: Periorbital edema enlarged towards the iris layer of the eye
  3. points: Periorbital edema covering the iris
  4. points: Severe periorbital edema covering the eyelid completely With this measurement tool, the periorbital edema status of all patients will be evaluated in terms of periorbital edema as stated above, and a score will be given by the researcher immediately after the patients come to the service from the operating room, at the 1st hour, 4th hour and 24th hour.
Right and left periorbital ecchymosis score | 1 hour after surgery
  Right and left periorbital ecchymosis; Right and left eyelids of all patients will be evaluated separately according to the following scale at the 1st, 4th and 24th hours, immediately after the patients come to the service from the operating room. Scoring diagram for ecchymosis; Grade 1, medial ecchymosis up to one-third of the lower and/or upper eyelid. Grade 2, ecchymosis up to the medial two-thirds of the lower and/or upper eyelid.
  3rd degree ecchymosis to the entire length of the lower and/or upper eyelid.
Right and left periorbital ecchymosis score | 4 hours after surgery
  Right and left periorbital ecchymosis; Right and left eyelids of all patients will be evaluated separately according to the following scale at the 1st, 4th and 24th hours, immediately after the patients come to the service from the operating room. Scoring diagram for ecchymosis; Grade 1, medial ecchymosis up to one-third of the lower and/or upper eyelid. Grade 2, ecchymosis up to the medial two-thirds of the lower and/or upper eyelid.
  3rd degree ecchymosis to the entire length of the lower and/or upper eyelid.
Right and left periorbital ecchymosis score | 24th hour after surgery
  Right and left periorbital ecchymosis; Right and left eyelids of all patients will be evaluated separately according to the following scale at the 1st, 4th and 24th hours, immediately after the patients come to the service from the operating room. Scoring diagram for ecchymosis; Grade 1, medial ecchymosis up to one-third of the lower and/or upper eyelid. Grade 2, ecchymosis up to the medial two-thirds of the lower and/or upper eyelid.
  3rd degree ecchymosis to the entire length of the lower and/or upper eyelid.

SECONDARY OUTCOMES:
Monitoring the change in fever | 1 hour after surgery 4 hours after surgery 24th hour after surgery
  Vital signs (fever) will be monitored every fifteen minutes in the first hour after the surgery, every thirty minutes in the next hour, and hourly thereafter.
Monitoring the change in systolic blood pressure | 1 hour after surgery 4 hours after surgery 24th hour after surgery
  Vital signs (systolic blood pressure) will be monitored every fifteen minutes in the first hour after the surgery, every thirty minutes in the next hour, and hourly thereafter.
Monitoring the change in diastolic blood pressure | 1 hour after surgery 4 hours after surgery 24th hour after surgery
  Vital signs (diastolic blood pressure) will be monitored every fifteen minutes in the first hour after the surgery, every thirty minutes in the next hour, and hourly thereafter.
Monitoring the change in pulse | 1 hour after surgery 4 hours after surgery 24th hour after surgery
  Vital signs (pulse) will be monitored every fifteen minutes in the first hour after the surgery, every thirty minutes in the next hour, and hourly thereafter.
Monitoring the change in oxygen saturation | 1 hour after surgery 4 hours after surgery 24th hour after surgery
  The change in the oxygen saturation values of the patients will be followed by noninvasive peripheral pulse oximetry.The patient's oxygen saturation value will be monitored every 4 hours, unlike the routine treatment and follow-up hours of the hospital. The saturation value will not be measured while the patient is asleep. A questionnaire will be applied to the patient to evaluate the patient's breathing in the morning after the surgery.
Richard's Campbell Sleep Scale | 1 hour after surgery 4 hours after surgery 24th hour after surgery
  It is a scale consisting of 6 items. These 6 items evaluate the depth of night sleep, the time to fall asleep, the frequency of waking up, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Evaluation of the scale, on the other hand, is that the score between 0-25 is "very bad sleep", and the score between "76-100" is "very good sleep". As the score of the scale increases, the sleep quality of the patients also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Şevval Polat, Principal Investigator — Uzunmehmet chest and occupational diseases hospital
Locations (1):
- Zonguldak Ataturk State Hospital, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No